CLINICAL TRIAL: NCT01278251
Title: Functional Review of Distal Biceps Re-Insertion
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Allegheny General Hospital
Other Study IDs: RC-4556
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Distal Biceps Ruptures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Endobutton
  Interventions: Procedure: Distal Biceps Re-Insertion

INTERVENTIONS:
Procedure: Distal Biceps Re-Insertion

SUMMARY:
This study seeks to test the hypothesis that endobutton repair of the ruptured distal biceps successfully restores elbow function.

ELIGIBILITY:
Inclusion Criteria:

* primary distal biceps repair with endobutton
* at least two years from date of surgery

Exclusion Criteria:

* any ipsilateral wrist, forearm, or elbow condition
* any contraindication to having an MRI

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have received primary distal biceps repair by Dr. Schmidt.
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Allegheny Imaging of McCandless, Pittsburgh, Pennsylvania, United States